CLINICAL TRIAL: NCT01274585
Title: Does Percutaneous Tibial Nerve Stimulation (PTNS) Improve Outcomes in Patients Presenting With Fecal Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to low recruitment rates
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Liliana Bordeianou, Colorectal Surgeon, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGH2010-P-000239
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No active treatment (Sham Comparator)
  Interventions: Device: Posterior tibial nerve stimulation
- stimulation/treatment (Experimental)
  Interventions: Device: Posterior tibial nerve stimulation (PTNS)

INTERVENTIONS:
Device: Posterior tibial nerve stimulation (PTNS) — Stimulation using PTNS device for 30 minutes weekly for 12 weeks
  Other Names: Urgent PC
  Arms: stimulation/treatment
Device: Posterior tibial nerve stimulation — Sham needle placement without active PTNS device for 30 minutes weekly for 12 weeks
  Arms: No active treatment

SUMMARY:
The primary objective of this study is to determine whether Percutaneous Tibial Nerve Stimulation (PTNS), a minimally invasive, simple, cost effective, and outpatient treatment of patients with urinary incontinence, can also be used to treat fecal incontinence. Specifically, the primary endpoint of this study is to determine, in a randomized controlled patient blinded study, whether PTNS decrease the episodes of fecal incontinence by 50% in the patients treated with PTNS when compared to placebo as documented by a 2 week patient bowel diary after treatment.

The investigators secondary endpoints will consist of measurements of the impact of PTNS on the severity of incontinence (defined as a decrease in the mean Fecal Incontinence Severity Index (FISI) score ), as well as on the patient quality of life factors related to fecal incontinence (defined as a decrease in the mean Fecal Incontinence Quality of Life (FIQoL) scale).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to provide informed consent
* Has severe fecal incontinence (defined as weekly episodes of incontinence of mucus, liquid or solid stool)
* Available to present for weekly treatments
* Available for follow-up at 3, 6, and 12 months

Exclusion Criteria:

1. Severe cardiopulmonary disease
2. Lesion of the Tibial Nerve
3. Use of a cardiac pacemaker or implantable defibrillator
4. History of inflammatory bowel disease
5. Active anal fissure, fistula, or abscess
6. Active rectal bleeding which has not been evaluated with appropriate testing, such as colonoscopy
7. Has a sphincter injury that needs sphincteroplasty
8. Wants to pursue aggressive surgical therapy with a colostomy or an artificial bowel sphincter
9. Severe distal venous insufficiency
10. Uncontrolled diabetes with peripheral nerve involvement
11. Immunosuppression
12. Pregnant or planning on becoming pregnant during treatment
13. Patients prone to bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Bordeianou, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Active Treatment | Stimulation/Treatment
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Active Treatment | Stimulation/Treatment | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 50 [33 to 66] | 69 [63 to 74] | 61 [33 to 74]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Fecal Incontinence
Description: Patient kept 2 week bowel diary after completion of treatment. Bowel diary were collected to assess frequency of fecal incontinence in the two week span.
Time Frame: Diary kept for 14 days following treatment
Measure: Mean (Full Range); unit: number of accidents
Arm/Group | No Active Treatment | Stimulation/Treatment
Number analyzed (Participants) | 2 | 3
number of accidents | 7.5 [2 to 13] | 33 [3 to 77]

2. Secondary Outcome: Change in Fecal Incontinence Severity Index (FISI) Score
Description: Fecal Incontinence Severity Index (FISI) is a tool used to stratify severity of fecal incontinence in the subjects. The range of score is from 0 to 61 where the higher score correlates with more severe symptoms of incontinence.
Time Frame: 12 weeks
Population: Only 4 of the 5 subjects completed questionnaires at the completion of the trial. Therefore, these were the only subjects included in analysis.
Measure: Mean (Full Range); unit: mean score
Arm/Group | No Active Treatment | Stimulation/Treatment
Number analyzed (Participants) | 2 | 2
mean score | 6 [5 to 7] | .5 [0 to 1]

3. Secondary Outcome: Change in Fecal Incontinence Quality of Life (FIQoL) Score
Description: The Fecal incontinence Quality of Life (FIQoL) score evaluates how fecal incontinence impacts the subjects quality of life. The scale ranges from 37 to 159 where the higher the score, the better the quality of life associated with symptoms.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Full Range); unit: mean score
Arm/Group | No Active Treatment | Stimulation/Treatment
Number analyzed (Participants) | 2 | 2
mean score | 11.5 [7 to 16] | 6.5 [2 to 11]

ADVERSE EVENTS:
Arm/Group | No Active Treatment | Stimulation/Treatment
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Active Treatment (N=2) | Stimulation/Treatment (N=3)
pain at needle site (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — pain when needle was inserted- resolved with removal of needle
hematoma at needle site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — small hematoma at needle site- found at following visit and resolved within 2 weeks
tingling in lower back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — tingling in back after procedure- resolved spontaneously prior to leaving clinic
abdominal cramping (Gastrointestinal disorders) | 1 (1) | 0 (0) — abdominal cramping after treatment. resolved spontaneously prior to leaving clinic
numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — subject had numbness after needle was removed. after moving around, resolved without further ill affects
GI bug (Gastrointestinal disorders) | 0 (0) | 2 (2) — subject reported 24 hour GI infection between treatments-resolved spontaneously without intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes